CLINICAL TRIAL: NCT06874920
Title: Outcomes of Empiric Antibiotic Treatment Based on Hospital Cumulative Antibiograms in Solid Organ Transplant Recipients with Bacteraemia: a Retrospective Single-centre Study (OPTIMIST Study)
Brief Title: Outcomes of Empiric Antibiotic Therapy Based on Hospital Antibiograms in Organ Transplant Recipients with Bacteraemia
Status: Enrolling by invitation | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Andrea Lombardi, Professor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 5392_20.11.2024_P_bis
Record Dates: First submitted 2025-02-06; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Bacteremia; Transplant Recipient
Keywords: Hospital cumulative antibiogram; Solid organ transplant; Bloodstream infections
MeSH Terms: conditions — Bacteremia; Sepsis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who was prescribed an empiric antibiotic therapy with OAS < 90%
  Interventions: Other: No intervention (observational study)
- Patients who was prescribed an empiric antibiotic therapy with OAS ≥ 90%
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
The purpose of this observational study is to examine how using the hospital cumulative antibiogram to guide empirical antibiotic therapy affects outcomes in patients with bloodstream infections who have undergone solid organ transplants. The key question is: does the use of a hospital cumulative antibiogram reduce mortality and improve outcomes in these patients?

DETAILED DESCRIPTION:
Sepsis is a critical condition responsible for more than 750,000 hospitalisations and 200,000 deaths annually in the US. Severe sepsis remains a leading cause of death worldwide, with in-hospital mortality ranging from 12% to 26% in the US. An early and appropriate antimicrobial therapy in sepsis leads to a decreased progression to septic shock and death. However, physicians are often unaware of microbiological results when confronting sepsis; moreover, adopting a broad spectrum antibiotic therapy can lead to multiple adverse events. Therefore, a good balance between antibiotic efficacy and the consequence of indiscriminate use of broad-spectrum antibiotics is necessary, particularly for immunocompromised individuals at a higher risk of severe sepsis. Different studies have addressed choosing adequate empiric antibiotic in sepsis: multivariable models using readily available epidemiologic factors to predict antimicrobial susceptibility and clinical decision tree to estimate multi-drug resistance (MDR) infections have been developed to help clinicians. Moreover, hospital cumulative antibiograms have been created to identify the most common sensitivity profile for every bacterium.

In this study we will analyse the potential role of hospital cumulative antibiograms in the outcome of solid organ transplant (SOT) recipients with bacteraemia. In particular, the primary objective of the study is to assess the 15-days mortality of SOT recipients with bacteraemia according to the treatment administered referred to overall antimicrobial susceptibility (OAS), while the secondary objectives of the study are to assess the 30-days mortality, the in-hospital mortality, the length of in-hospital, the ICU admission, and the length of Intensive Care Unit (ICU) stay in these patients. Moreover, we will also assess the frequency of empiric therapy change at antibiogram availability, and we will describe the reasons for empiric therapy change.

We will conduct a retrospective single-centre cohort study to investigate the effect of empiric antibiotic treatment according to OAS on outcomes of the target population composed by SOT recipients transplanted in our Centre who were hospitalized at Fondazione IRCCS Ca' Granda Policlinico of Milano from 01/01/2015 to 31/12/2023 and developed monomicrobial bloodstream infection (BSI) due to Acinetobacter baumannii, Enterobacter spp., Enterococcus faecalis, Enterococcus faecium, Escherichia coli, Klebsiella pneumoniae, Klebsiella other-than pneumoniae, Proteus mirabilis, Pseudomonas aeruginosa, Serratia marcescens, Staphylococcus aureus, Staphylococcus lugdunensis, and Streptococcus spp.

Patients will be divided into two groups according to the overall antimicrobial susceptibility of the empiric antibiotic therapy prescribed based on hospital cumulative antibiograms:

* Patients who have been prescribed an empiric therapy with OAS < 90%;
* Patients who have been prescribed an empiric therapy with OAS ≥ 90%. Hospital cumulative antibiograms of the years included in the study are already available for the following temporal periods: 2014, 2015, 2016, 2017, 2018, 2019, 2020, 2021, 2022 and 2023. OAS is defined as the ratio of strains of a pathogen which are sensitive to an antibiotic regimen referred to all the strain of this pathogen identified.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Being SOT
* Monomicrobial bloodstream infection due to Acinetobacter baumannii, Enterobacter spp., Enterococcus faecalis, Enterococcus faecium, Escherichia coli, Klebsiella pneumoniae, Klebsiella other-than pneumoniae, Proteus mirabilis, Pseudomonas aeruginosa, Serratia marcescens, Staphylococcus aureus, Staphylococcus lugdunensis, and Streptococcus spp.
* Hospitalization in Fondazione IRCCS Cà Granda Policlinico of Milano from 2015 to 2023.

Exclusion Criteria:

* Antibiotic therapy administration outside 48h before-after blood culture collection.
* Polymicrobial bloodstream infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Solid organ transplant recipients with bloodstream infections.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
15-days mortality | 15 days from bloodstream infection

SECONDARY OUTCOMES:
30-days mortality | 30 days from bloodstream infection
In-hospital mortality | Up to 24 weeks
  From bloodstream infection to hospital discharge
Lenght of hospital stay | Up to 24 weeks
  From hospital admission to hospital discharge
ICU admission | Up to 24 weeks
  From bloodstream infection to hospital discharge
Lenght of ICU stay | Up to 24 weeks
  From ICU admission to ICU discharge
Frequency of empiric therapy change at antibiogram availability | Up to five days
  From empiric antibiotic therapy prescription to targeted antibiotic therapy prescription
Reason for empiric antibiotic change | From empiric antibiotic therapy prescription to targeted antibiotic therapy prescription at 5 days
  Change from empiric to targeted antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided